CLINICAL TRIAL: NCT02504346
Title: AZD9291, an Irreversible EGFR-TKI, in Relapsed EGFR-mutated Non-small Cell Lung Cancer Patients Previously Treated With an EGFR-TKI, Coupled to Extensive Translational Studies
Acronym: TREM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Odd Terje Brustugun, Senior consultant, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/10301
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Targeted Therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Non-randomized trial, all patients receive therapy - singel-arm
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291

SUMMARY:
Phase II, single-arm study to assess the safety and efficacy of AZD9291 (80 mg, orally, once daily) in second-line (or later) patients with EGFR mutation-positive, locally advanced or metastatic NSCLC, who have progressed following treatment with an approved epidermal growth factor tyrosine kinase inhibitor agent.

DETAILED DESCRIPTION:
This is a phase II, single-arm study to assess the safety and efficacy of AZD9291 (80 mg, orally, once daily) in second-line (or later) patients with EGFR mutation-positive, locally advanced or metastatic NSCLC, who have progressed following treatment with an approved epidermal growth factor tyrosine kinase inhibitor agent.

If feasible, subjects will have to provide a biopsy sample for molecular testing following confirmed disease progression on the most recent treatment regimen. A second biopsy will be sampled at progression on AZD9291, if feasible. Liquid biopsies will be sampled throughout the treatment period.

Subjects should continue on study treatment until RECIST 1.1-defined progression or until a treatment discontinuation criterion is met. There is no maximum duration of treatment as subjects may continue to receive investigational product beyond RECIST 1.1 defined progression as long as they are continuing to show clinical benefit, as judged by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent.
2. Age > 18 years.
3. Histologically or cytologically documented locally advanced or metastatic NSCLC not amenable to curative surgery or radiotherapy.
4. Radiological disease progression following at least one prior EGFR TKI.
5. Documented EGFR mutation known to be associated with EGFR TKI sensitivity (also including T790M).
6. ECOG status 0-2 and a minimum life expectancy of 12 weeks.
7. At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline according to RECIST 1.1.
8. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
9. Male subjects must be willing to use barrier contraception.

   -

Exclusion Criteria:

* 1. Treatment with an EGFR-TKI within 8 days or approximately 5x half-life, whichever is the longer, of the first dose of study treatment.

  2. Treatment with cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days or approximately 5x half-life, whichever is the longer, of the first dose of study treatment.

  3. Previous treatment with AZD9291, or another EGFR TKI with similar profile, e.g. CO-1686 4. Major surgery within 4 weeks of inclusion 5. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of inclusion 6. Subjects currently receiving (or unable to stop using) potent inhibitors or inducers of CYP3A4 7. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 (with the exception of alopecia grade 2) at the time of starting study treatment.

  8. Spinal cord compression or brain metastases unless asymptomatic and on stable steroid dosage for at least 2 weeks prior to start of study treatment.

  9. Any evidence of severe or uncontrolled systemic diseases which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.

  10. Gastrointestinal conditions incompatible with swallowing or precluding absorption of AZD9291.

  11. Exclude based on any of the following cardiac criteria:
* Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval 12. Current or previous significant interstitial lung disease or radiation pneumonitis 13. Absolute neutrophil count < 1.5 x 109/L 14. Platelet count < 100 x 109/L 15. Haemoglobin < 80 g/L 16. Alanine aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases 17. Aspartate aminotransferase (AST) > 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases 18. Total bilirubin > 1.5 times ULN if no liver metastases or > 3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases 19. Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 ml/min (measured or calculated by Cockcroft and Gault equation), 20. History of hypersensitivity of AZD9291 (or drugs with a similar chemical structure or class.

  21. Women who are pregnant or breast-feeding, or have a positive (urine or serum) pregnancy test prior to study entry 22. Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 weeks
  Measured by RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (7):
- Herlev Hospital, Copenhagen, Denmark
- Oulu University Hospital, Oulu, Finland
- National Cancer Institute, Vilnius, Lithuania
- Norway (3):
  - Drammen Hospital - Vestre Viken HF, Drammen
  - Norwegian Radium Hospital, Oslo
  - St Olavs hospital, Trondheim
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Eide IJZ, Helland A, Ekman S, Mellemgaard A, Hansen KH, Cicenas S, Koivunen J, Gronberg BH, Brustugun OT. Osimertinib in T790M-positive and -negative patients with EGFR-mutated advanced non-small cell lung cancer (the TREM-study). Lung Cancer. 2020 May;143:27-35. doi: 10.1016/j.lungcan.2020.03.009. Epub 2020 Mar 12. PMID 32200138